CLINICAL TRIAL: NCT00830271
Title: Pilot Study of Vicryl Plus and Monocryl Plus in Breast Surgery
Brief Title: Vicryl Plus and Monocryl Plus in Breast Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiff and Vale University Health Board (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C624/07
Record Dates: First submitted 2009-01-21; First posted 2009-01-27 (Estimated); Last update posted 2020-01-30 (Actual); Status verified 2009-01

CONDITIONS: Breast Cancer Surgery
Keywords: surgical site infection; wound complications; suture; antiseptic; wound closure
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vicryl plus/Monocryl plus (Experimental): Vicryl plus and Monocryl plus is the active comparator arm. These are the "active" sutures, coated with triclosan antiseptic, being used in the closure of skin and subcutaneous tissues after breast cancer surgery.
  Interventions: Device: Vicryl plus and Monocryl plus
- vicryl/monocryl (Placebo Comparator): "Plain" Vicryl or Monocryl suture currently the standard which are not coated with triclosan, serve as the control.
  Interventions: Device: wound closure with Vicryl and Monocryl

INTERVENTIONS:
Device: Vicryl plus and Monocryl plus — closure of skin and subcutaneous tissues
  Arms: Vicryl plus/Monocryl plus
Device: wound closure with Vicryl and Monocryl — wound closure skin and subcutaneous tissues
  Arms: vicryl/monocryl

SUMMARY:
This is a randomised pilot study comparing conventional sutures (Vicryl and Monocryl) with antiseptic coated equivalents (Vicryl plus andf Monocryl plus) in elective breast surgery.

ELIGIBILITY:
Inclusion Criteria:

* All patients over 18 years old who attend the Cardiff and Vale NHS Trust for elective breast cancer surgery

Exclusion Criteria:

* patients unable to give consent or comply with follow up
* patients undergoing surgery for benign disease
* patients with inflammatory cancers or skin ulceration
* patients having neo-adjuvant chemotherapy or radiotherapy
* patients with known allergy to triclosan antiseptic
* patients with immune deficiency diseases

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2008-12; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
reduction of surgical site infection | 6-7 months

SECONDARY OUTCOMES:
estimation time in hospital and return to work numbers of haematomas and seromas | 6-9 months

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiff and Vale NHS Trust, Cardiff, Wales, United Kingdom